CLINICAL TRIAL: NCT02802345
Title: INSTAGE: A 24-week, Double-blind, Randomized, Parallel-group Study Evaluating the Efficacy and Safety of Oral Nintedanib Co-administered With Oral Sildenafil, Compared to Treatment With Nintedanib Alone, in Patients With Idiopathic Pulmonary Fibrosis (IPF) and Advanced Lung Function Impairment
Brief Title: Efficacy and Safety of Nintedanib Co-administered With Sildenafil in Idiopathic Pulmonary Fibrosis Patients With Advanced Lung Function Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.36; 2015-002619-14 (EudraCT Number)
Expanded Access: Available
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nintedanib + placebo matching sildenafil (Experimental)
  Interventions: Drug: Nintedanib; Drug: Placebo
- Nintedanib + Sildenafil (Active Comparator)
  Interventions: Drug: Nintedanib; Drug: Sildenafil

INTERVENTIONS:
Drug: Nintedanib
Drug: Placebo
  Arms: Nintedanib + placebo matching sildenafil
Drug: Sildenafil
  Arms: Nintedanib + Sildenafil

SUMMARY:
To assess efficacy and safety of concomitant treatment with nintedanib and sildenafil in Idiopathic Pulmonary Fibrosis (IPF) patients with advanced lung function impairment.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent consistent with International Conference on Harmonization-Good Clinical Practice and local laws, signed prior to any study procedures being performed (including any required washout);
* Male or female patients aged >= 40 years at visit 1;
* A clinical diagnosis of IPF within the last 6 years before visit 1, based upon the American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American thoracic Association 2011 guideline [P11-07084];
* Combination of high-resolution computed tomography (HRCT) pattern, and if available, surgical lung biopsy pattern consistent with a diagnosis of IPF as assessed by the investigator based on a HRCT scan performed within 18 months of visit 1;
* Carbon Monoxide Diffusion Capacity (corrected for Hb) less or equal to 35% predicted of normal at visit 1.

Exclusion criteria:

* Previous enrolment in this trial;
* Alanine Transaminase, Aspartate Transaminase > 1.5 fold upper limit of normal (ULN) at visit 1;
* Total bilirubin > 1.5 fold ULN at visit 1;
* Relevant airways obstruction (i.e. pre-bronchodilator Forced Expiratory Volume in 1 second/Forced Vital Capacity <0.7 at visit 1)
* History of myocardial infarction within 6 months of visit 1 or unstable angina within 1 month of visit 1
* Bleeding Risk:

  * Known genetic predisposition to bleeding;
  * Patients who require fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin, etc.) or high dose antiplatelet therapy;
  * History of haemorrhagic central nervous system (CNS) event within 12 months prior to visit 1;
  * History of haemoptysis or haematuria, active gastro-intestinal bleeding or ulcers and/or major injury or surgery within 3 months prior to visit 1;
  * International normalised ratio (INR) > 2 at visit 1;
  * Prothrombin time (PT) and activated partial thromboplastin time (aPTT) > 150% of institutional ULN at visit 1;
* Planned major surgery during the trial participation, including lung transplantation, major abdominal or major intestinal surgery;
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of visit 1;
* Creatinine clearance < 30 mL/min calculated by Cockcroft-Gault formula at visit 1;
* Presence of aortic stenosis (AS) per investigator judgement at visit 1;
* Severe chronic heart failure: defined by left ventricular ejection fraction (EF) < 25% per investigator judgement at visit 1;
* Presence of idiopathic hypertrophic subaortic stenosis (IHSS) per investigator judgement at visit 1;
* Second-degree or third-degree atrioventricular (AV) block on electrocardiogram (ECG) per investigator judgement at visit 1;
* Hypotension (systolic blood pressure [SBP] < 100 mm Hg or diastolic blood pressure [DBP] < 50 mm Hg) (symptomatic orthostatic hypotension) at visit 1;
* Uncontrolled systemic hypertension (SBP > 180 mmHg; or DBP > 100 mmHg) at visit 1;
* Known penile deformities or conditions (e.g., sickle cell anemia, multiple myeloma, leukemia) that may predispose to priapism;
* Retinitis pigmentosa;
* History of vision loss;
* History of nonarteritic ischemic optic neuropathy;
* Veno-occlusive disease;
* History of acute IPF exacerbation or respiratory infection within 8 weeks of visit 2.
* Treatment with nitrates, n-acetylcysteine, pirfenidone, azathioprine, cyclophosphamide, cyclosporine, prednisone >15 mg daily or >30 mg every 2 days OR equivalent dose of other oral corticosteroids as well as any investigational drug within 4 weeks of visit 2;
* Treatment with prostaglandins (e.g., epoprostenol, treprostinil), endothelin-1 antagonists (e.g., bosentan, sitaxsentan, ambrisentan), phosphodiesterase inhibitors (e.g., sildenafil, tadalafil, vardenafil) or a stimulator of guanylatcyclase (e.g.,riociguat) within 4 weeks of visit 2;
* Treatment with potent cytochrome CYP3A4 inhibitors such as ketoconazole, itraconazole and ritonavir within 4 weeks of visit 2;
* Supplementation with L-arginine and concurrent use of grapefruit juice or St John's wort within 4 weeks of visit 2;
* Treatment with the reduced dose of nintedanib (100 mg bid) within 4 weeks of visit 2; 27. Permanent discontinuation of nintedanib in the past due to adverse events considered drug-related;
* Known hypersensitivity or intolerance to nintedanib, sildenafil, galactose, peanut or soya or any other components of the study medication;
* A disease or condition which in the opinion of the investigator may interfere with testing procedures or put the patient at risk when participating in this trial;
* Alcohol or drug abuse which in the opinion of the treating physician would interfere with treatment;
* Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (85):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Assoc of Stamford, Stamford, Connecticut
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Michigan Clinical Research Unit, Ann Arbor, Michigan
  - Minnesota Lung Center, Minneapolis, Minnesota
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Research Solutions, Dayton, Ohio
  - Mercy Respiratory Specialist, Toledo, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Lowcountry Lung and Crit Care, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (3):
  - Ziekenhuis Netwerk Antwerpen (ZNA) - Campus Middelheim, Antwerp
  - ULB Hopital Erasme, Brussels
  - UZ Leuven, Leuven
- Canada (5):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre (Dalhousie University), Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
- France (8):
  - HOP Louis Pradel, Bron
  - HOP Calmette, Lille
  - HOP Nord, Marseille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - HOP Européen G. Pompidou, Paris
  - HOP Bichat, Paris
  - HOP Pontchaillou, Rennes
- Germany (8):
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Universitätsmedizin Greifswald, Greifswald
  - Medizinische Hochschule Hannover, Hanover
  - Lungenfachklinik Immenhausen, Immenhausen
  - Wissenschaftliches Institut Bethanien, Solingen
- India (5):
  - Sanjivani Superspeciality Hospital Pvt. Ltd., Ahmedabad
  - Care Institute Of Medical Sciences, Ahmedabad
  - Sri Bala Medical Centre & Hospitals, Coimbatore
  - Fortis Hospital, Kolkata
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune
- Italy (10):
  - Osp. Clin. SS. Anunziata, Chieti Scalo
  - Ospedale Colonnello D Avanzo, Foggia
  - Ospedale "G.B. Morgagni - L. Pierantoni" ausl forli, Forlì
  - Osp. S. Giuseppe Fatebenefratelli, Milan
  - Università di Modena e Reggio Emilia, Modena
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Az. Ospedaliera Universitaria Polic.Tor Vergata, Roma
  - Policlinico Gemelli, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - Ospedale Riuniti di Ancona, Torrette Di Ancona (Ancona)
- Japan (9):
  - Tosei General Hospital, Aichi, Seto
  - Kurume University Hospital, Fukuoka, Kurume
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Toho University Omori Medical Center, Tokyo, Ota-ku
- Mexico (4):
  - Nuevo Hospital Civil de Guadalajara DR. JUAN I. MENCHACA, Guadalajara
  - Centro Respiratorio de Mexico, México
  - Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas, México
  - Centro de Prevención y Rehabilitación de Enfermedades Pulmon, Monterrey
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (6):
  - Southmead Hospital, Bristol
  - Papworth Hospital, Cambridge
  - Ninewells Hospital & Medical School, Dundee, Scotland
  - Queen Elizabeth University Hospital, Glasgow
  - Northern General Hospital, Sheffield
  - South Tyneside District Hospital, Tyne and Wear

REFERENCES:
- [Derived] Richeldi L, Kolb M, Jouneau S, Wuyts WA, Schinzel B, Stowasser S, Quaresma M, Raghu G. Efficacy and safety of nintedanib in patients with advanced idiopathic pulmonary fibrosis. BMC Pulm Med. 2020 Jan 8;20(1):3. doi: 10.1186/s12890-019-1030-4. PMID 31914963
- [Derived] Behr J, Kolb M, Song JW, Luppi F, Schinzel B, Stowasser S, Quaresma M, Martinez FJ. Nintedanib and Sildenafil in Patients with Idiopathic Pulmonary Fibrosis and Right Heart Dysfunction. A Prespecified Subgroup Analysis of a Double-Blind Randomized Clinical Trial (INSTAGE). Am J Respir Crit Care Med. 2019 Dec 15;200(12):1505-1512. doi: 10.1164/rccm.201903-0488OC. PMID 31365829
- [Derived] Kolb M, Raghu G, Wells AU, Behr J, Richeldi L, Schinzel B, Quaresma M, Stowasser S, Martinez FJ; INSTAGE Investigators. Nintedanib plus Sildenafil in Patients with Idiopathic Pulmonary Fibrosis. N Engl J Med. 2018 Nov 1;379(18):1722-1731. doi: 10.1056/NEJMoa1811737. Epub 2018 Sep 15. PMID 30220235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, double-blind, parallel design comparison of nintedanib 150 milligram (mg) twice daily (bid) and sildenafil 20 mg three times a day (tid) to nintedanib 150 mg bid and placebo matching sildenafil tid administered orally over 24 weeks.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all patients met all inclusion/exclusion criteria. Patients were not to be randomized to trial if any one of the specific entry criteria were not met.
Groups:
- Nintedanib+Placebo: Patients administered 150 milligram (mg) soft gelatine capsule orally twice daily (bid), with a possibility of dose reduction to 100 mg capsule bid along with placebo matching to Sildenafil for 24 weeks.
- Nintedanib+Sildenafil: Patients administered 150 milligram (mg) soft gelatine capsule orally twice daily (bid), with a possibility of dose reduction to 100 mg capsule bid along with 20 mg thrice daily (tid) Sildenafil for 24 weeks.
Period: Overall Study
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil
Started | 136 | 138
Treated | 136 | 137
Completed (Completed Nintedanib treatment) | 104 | 108
Not Completed | 32 | 30
Not completed — Not Treated | 0 | 1
Not completed — Adverse Event | 28 | 20
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Other than listed | 1 | 5

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): TS included all patients who were randomised to a treatment group and received at least one dose of randomised study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil | Total
Number analyzed (Participants) | 136 | 137 | 273
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set (TS): TS included all patients who were randomised to a treatment group and received at least one dose of randomised study medication.
  Years | 70.0 (7.9) | 70.3 (8.6) | 70.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set (TS): TS included all patients who were randomised to a treatment group and received at least one dose of randomised study medication.
  Participants
    Female | 30 | 27 | 57
    Male | 106 | 110 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set (TS): TS included all patients who were randomised to a treatment group and received at least one dose of randomised study medication.
  Participants
    Hispanic or Latino | 15 | 23 | 38
    Not Hispanic or Latino | 121 | 114 | 235
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated Set (TS): TS included all patients who were randomised to a treatment group and received at least one dose of randomised study medication.
  Participants
    American Indian or Alaska Native | 2 | 3 | 5
    Asian | 39 | 30 | 69
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 95 | 103 | 198
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Total Score at Week 12
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life). Scores are calculated for three domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A minimum change in score of 4 units was established as clinically relevant after patient and clinician testing. Scores range from 0 to 100, with higher scores indicating more limitations. The mean and standard error presented are actually adjusted mean for change from baseline and its standard error.
Time Frame: Baseline and week 12
Population: TS
Measure: Mean (Standard Error); unit: Unit on scale
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil
Number analyzed (Participants) | 133 | 132
Unit on scale | -0.77 (1.009) | -1.28 (1.013)
Statistical Analysis 1: Comparison: Nintedanib+Placebo vs Nintedanib+Sildenafil; Mixed Model for Repeated Measures (MMRM) included fixed effects for treatment, visit, presence of any echocardiographic signs, baseline SGRQ total score as covariate, treatment-by-visit and baseline SGRQ total score-by-visit interaction terms using an unstructured covariance matrix. No imputation was planned. Data collected after Visit 5 (planned 12 weeks after start of study treatment) were not used for this analysis; Test type: Superiority; p = 0.7191, Mixed Model for Repeated Measures (MMRM); The Roger- Kenward approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = -0.52, 95% CI 2-sided [-3.33 to 2.30], Standard Error of Mean 1.431 — Adjusted mean difference (Nintedanib +placebo vs Nintedanib+sildenafil) is based on all analyzed patients in the model (not only patients with a measurement at baseline and at 12 weeks); H0: There is no difference in the mean change from baseline in SGRQ total score at Week 12 between treatment with nintedanib co-administered with sildenafil and treatment with nintedanib alone. Ha: There is a difference in the mean change from baseline in SGRQ total score at Week 12 between treatment with nintedanib co-administered with sildenafil and treatment with nintedanib alone

2. Secondary Outcome: Change From Baseline in Dyspnoea Using the University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ) at Week 12
Description: The UCSD SOBQ is a 24-item questionnaire developed to measure breathlessness on a scale between zero and five where 0 is not at all breathless and 5 is maximally breathless or too breathless to do the activity. The mean and standard error presented for descriptive statistics are actually adjusted mean for change from baseline and its standard error.
Time Frame: Baseline and week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil
Number analyzed (Participants) | 122 | 120
Unit on scale | 4.40 (1.529) | 1.46 (1.575)
Statistical Analysis 1: Comparison: Nintedanib+Placebo vs Nintedanib+Sildenafil; Mixed Model for Repeated Measures (MMRM) included fixed effects for treatment, visit, presence of any echocardiographic signs, baseline UCSD SOBQ total score as covariate, treatment-by-visit and baseline UCSD SOBQ total score-by-visit interaction terms using an unstructured covariance matrix. No imputation was planned. Data collected after Visit 5 (planned 12 weeks after start of study treatment) were not used for this analysis; Test type: Superiority; p = 0.1823, Mixed Model for Repeated Measures (MMRM); The Roger- Kenward approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = -2.94, 95% CI 2-sided [-7.27 to 1.39], Standard Error of Mean 2.198 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in SGRQ Total Score at Week 24
Description: The SGRQ is a 50-item questionnaire developed to measure health status (quality of life). Scores are calculated for three domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A minimum change in score of 4 units was established as clinically relevant after patient and clinician testing. The mean and standard error presented for descriptive statistics are actually adjusted mean for change from baseline and its standard error.
Time Frame: Baseline and week 24
Population: TS
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil
Number analyzed (Participants) | 133 | 132
Unit on scale | 2.42 (1.158) | 0.23 (1.148)
Statistical Analysis 1: Comparison: Nintedanib+Placebo vs Nintedanib+Sildenafil; Mixed Model for Repeated Measures (MMRM) included fixed effects for treatment, visit, presence of any echocardiographic signs, baseline SGRQ total score as covariate, treatment-by-visit and baseline SGRQ total score-by-visit interaction terms using an unstructured covariance matrix. No imputation was planned; Test type: Superiority; p = 0.1809, Mixed Model for Repeated Measures (MMRM); The Roger- Kenward approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = -2.19, 95% CI 2-sided [-5.40 to 1.02], Standard Error of Mean 1.631 — Adjusted mean difference (Nintedanib +placebo vs Nintedanib+sildenafil) is based on all analyzed patients in the model (not only patients with a measurement at baseline and at 24 weeks)

4. Secondary Outcome: Change From Baseline in Dyspnoea Using UCSD SOBQ at Week 24
Description: The UCSD SOBQ is a 24-item questionnaire developed to to measure breathlessness on a scale between zero and five where 0 is not at all breathless and 5 is maximally breathless or too breathless to do the activity. The mean and standard error presented for descriptive statistics are actually adjusted mean for change from baseline and its standard error.
Time Frame: Baseline and week 24
Population: TS
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil
Number analyzed (Participants) | 124 | 123
Unit on scale | 6.85 (1.791) | 4.44 (1.779)
Statistical Analysis 1: Comparison: Nintedanib+Placebo vs Nintedanib+Sildenafil; Mixed Model for Repeated Measures (MMRM) included fixed effects for treatment, visit, presence of any echocardiographic signs, baseline UCSD SOBQ total score as covariate, treatment-by-visit and baseline UCSD SOBQ total score-by-visit interaction terms using an unstructured covariance matrix. No imputation was planned; Test type: Superiority; p = 0.3421, Mixed Model for Repeated Measures (MMRM); The Roger- Kenward approximation was used to estimate denominator degrees of freedom; Adjusted mean difference = -2.41, 95% CI 2-sided [-7.39 to 2.58], Standard Error of Mean 2.529 — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Percentage of Patients With On-treatment Serious Adverse Events (SAE) From Baseline to Week 24
Description: Percentage of patients with on-treatment serious adverse events (SAE) from baseline to Week 24 is presented.
Time Frame: Baseline and week 24
Population: TS
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil
Number analyzed (Participants) | 136 | 137
Percentage of participants (%) | 32.4 | 27.0
Statistical Analysis 1: Comparison: Nintedanib+Placebo vs Nintedanib+Sildenafil; Relative risk, Comparison of treatment groups is calculated by Cochran-Mantel-Haenszel test adjusting for the categorical covariate presence of any echocardiographic signs indicative of right heart dysfunction (yes/no), adjusted Mantel-Haenszel type risk ratios and risk differences with 95% confidence are presented; Test type: Superiority; Percentage ratio (%) = 0.83, 95% CI 2-sided [0.58 to 1.20] — Within strata confidence limits are calculated according to Wald. Percentage ratio = (% of Nintedanib+sildenafil) / (% of Nintedanib+placebo)
Statistical Analysis 2: Comparison: Nintedanib+Placebo vs Nintedanib+Sildenafil; Risk difference, Comparison of treatment groups is calculated by Cochran-Mantel-Haenszel test adjusting for the categorical covariate presence of any echocardiographic signs indicative of right heart dysfunction (yes/no), adjusted Mantel-Haenszel type risk ratios and risk differences with 95% confidence are presented; Test type: Superiority; p = 0.334, Cochran-Mantel-Haenszel; Percentage difference (%) = -5.37, 95% CI 2-sided [-16.25 to 5.52] — Within strata confidence limits are calculated according to Wald. Percentage difference = (% of Nintedanib+sildenafil) - (% of Nintedanib+placebo)

ADVERSE EVENTS:
Time Frame: From first drug administration to 28 days after the last trial medication administration, 227 days.
Arm/Group | Nintedanib+Placebo | Nintedanib+Sildenafil
All-Cause Mortality (participants affected / at risk) | 12/136 | 12/137
Serious Adverse Events (participants affected / at risk) | 44/136 | 37/137
Other Adverse Events (participants affected / at risk) | 113/136 | 118/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib+Placebo (N=136) | Nintedanib+Sildenafil (N=137)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 5
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1
Eosinophil percentage increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib+Placebo (N=136) | Nintedanib+Sildenafil (N=137)
Abdominal pain (Gastrointestinal disorders) | 9 | 4
Abdominal pain upper (Gastrointestinal disorders) | 7 | 6
Constipation (Gastrointestinal disorders) | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 66 | 79
Dyspepsia (Gastrointestinal disorders) | 4 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 7
Nausea (Gastrointestinal disorders) | 14 | 22
Vomiting (Gastrointestinal disorders) | 9 | 19
Asthenia (General disorders) | 7 | 6
Fatigue (General disorders) | 6 | 7
Oedema peripheral (General disorders) | 6 | 7
Pyrexia (General disorders) | 9 | 6
Bronchitis (Infections and infestations) | 4 | 12
Influenza (Infections and infestations) | 7 | 4
Nasopharyngitis (Infections and infestations) | 8 | 9
Respiratory tract infection (Infections and infestations) | 4 | 8
Alanine aminotransferase increased (Investigations) | 8 | 8
Aspartate aminotransferase increased (Investigations) | 7 | 5
C-reactive protein increased (Investigations) | 7 | 6
Gamma-glutamyltransferase increased (Investigations) | 7 | 7
Weight decreased (Investigations) | 12 | 7
Decreased appetite (Metabolism and nutrition disorders) | 23 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Dizziness (Nervous system disorders) | 8 | 6
Headache (Nervous system disorders) | 10 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT02802345/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT02802345/SAP_001.pdf